CLINICAL TRIAL: NCT06715644
Title: ROX Index Versus MROX Index to Predict Treatment Outcome for High Flow Nasal Cannula And/or Noninvasive Ventilation in Patients with Respiratory Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ramadan Abd el rahman Ibraheim, resident doctor at Chest Diseases and Tuberculosis department Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: ROX mROX HFNC RF
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Failure
Keywords: ROX index; mROX index; high flow nasal cannula; noninvasive ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: patients with respiratory failure treated with high flow nasal cannula
- group 2: patients with respiratory failure treated with noninvasive ventilation in

SUMMARY:
One of managing steps in respiratory failure is high flow nasal cannula (HFNC), but the exact time to turn to invasive machine ventilation (IMV) is necessarily being determined. Respiratory rate and oxygenation (ROX) index, defined as the ratio of oxygen saturation as measured by pulse oximetry (SO2)/ FiO2 to respiratory rate (RR), is used to determine when to intubate the patients who are on HFNC and prevent the delayed intubation. Modified Respiratory rate and oxygenation (mROX), defined as (PaO2/ FiO2) / respiratory rate, is also used to point the time of intubation in case HFNC of patients with respiratory failure . The diagnostic and prognostic accuracy of both parameters are reported in previous papers, but the preference of them is under research. In this study, we aim to observe and compare the diagnostic accuracy between ROX and mROX in determine the time of invasive mechanical ventilation.

DETAILED DESCRIPTION:
Respiratory Failure (RF) is a condition where there's insufficient oxygenation in the body tissue, whether acute, chronic or acute on chronic; occurring due to decreased oxygen or excessive carbon-dioxide in the blood . There are four types of respiratory failure; Hypoxemic respiratory failure (Type1), hypercapnic respiratory failure (Type2), ) . Causes of RF are varied and accounted for any abnormality related upper respiratory tract, lower respiratory tract, central and peripheral nervous system or muscles of respiration . However, in the last three decades, the most common causes of RF is acute myocardial infarction (AMI), acute respiratory distress syndrome (ARDS), RF related to corona virus (Covid-19) and acute exacerbation of chronic obstructive lung disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sex aged between 18 to 80 years
* Patient diagnosed with acute type 1or 2 or chronic type 1or 2 respiratory failure.
* Patient for chest ICU admission
* Patient for HFNC and/ or Noninvasive mechanical ventilation.

Exclusion Criteria:

* Pediatric patients
* Pregnant females
* Patients who are for intubation on ICU admissionc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with acute type 1or 2 or chronic type 1or 2 respiratory failure.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of ROX in determine the time of invasive mechanical ventilation. | baseline
  Sensitivity and Specificity in determine the time of invasive mechanical ventilation.

SECONDARY OUTCOMES:
diagnostic accuracy mROX index in determine the time of invasive mechanical ventilation. | baseline
  Sensitivity and Specificity of mROX index in determine the time of invasive mechanical ventilation.

IPD SHARING:
Plan to Share IPD: Undecided